CLINICAL TRIAL: NCT01257711
Title: A Prospective Randomised Study Comparing Billroth II With Roux-en-Y Reconstruction After Radical Distal Subtotal Gastrectomy for Gastric Cancer
Brief Title: A Study Comparing Billroth II With Roux-en-Y Reconstruction for Gastric Cancer
Acronym: SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: Tan Tock Seng Hospital (Other); Changi General Hospital (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Asim Shabbir, Doctor, National Healthcare Group, Singapore
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B/08/333
Record Dates: First submitted 2010-06-08; First posted 2010-12-10 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Gastric Cancer; Stomach Cancer; Gastrectomy
Keywords: Gastric Cancer; Gastrectomy; Billroth 2; Roux-en-Y
MeSH Terms: conditions — Stomach Neoplasms | interventions — Anastomosis, Roux-en-Y; Gastroenterostomy; Plastic Surgery Procedures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Billroth II reconstruction (Other): Following Radical Distal Subtotal Gastrectomy, patient will be randomised to restore the continuity of the intestine with the stomach using Billroth II reconstruction.
  Interventions: Procedure: Roux-en-Y or Billroth II
- Roux-en-Y reconstruction (Other): Following Radical Distal Subtotal Gastrectomy, patient will be randomised to restore the continuity of the intestine with the stomach using Roux-en-Y reconstruction.
  Interventions: Procedure: Roux-en-Y or Billroth II

INTERVENTIONS:
Procedure: Roux-en-Y or Billroth II — Roux-en-Y had fewer problems related to reflux of bile but a higher incidence of stasis in the Roux limb resulting in longer hospital stay. Some surgeon avoids doing Roux-en-Y is a triad of post operative symptoms including abdominal pain, vomiting and nausea called Roux-en-Y loop syndrome. Billroth II reconstruction is a simpler operation with only one anastomosis and faster operating time. This has implications while managing gastric cancer patients who may be malnourished and a simpler procedure may have lesser risk of complications and yield better outcomes. Billroth II has increased reflux associated problem like esophagitis and gastritis, risk of afferent loop and dumping syndrome. Long term nutritional outcomes are similar for both procedures.
  Other Names: Reconstruction

SUMMARY:
Both Billroth II and Roux en Y are acceptable techniques of reconstruction after subtotal gastrectomy, however the debate one which is better remains unanswered. The aim of this study is to compare Billroth II and Roux en Y reconstruction techniques after radical distal subtotal gastrectomy for gastric cancer in terms of postoperative outcomes and quality of life. The investigators hypothesize that Roux en Y will have lesser gastrointestinal symptoms and reflux problems when compared to Billroth II reconstruction. Patients with resectable gastric cancer meeting the inclusion criteria will be consented and enrolled. Data on demographics, nutrition, gastrointestinal symptoms, and quality of life will be collected. They will be randomized after completion of distal subtotal gastrectomy to under go either Roux en Y or Billroth II reconstruction. Surgery data will be collected post-operatively.

At 6 months follow up a repeat nutritional assessment using clinical and biochemical parameters will be carried out. The biochemical markers are part of routine follow up. The final assessment will be at the one year post surgery visit when by interview using EORTC 30 questionnaire quality of life data, gastrointestinal symptoms and nutritional assessment and surgery data for recurrence will be repeated. At one year patients will also have upper gastrointestinal endoscopy, which is part of routine follow up. At endoscopy stump gastritis will be graded and esophageal reflux assessed as per Los Angeles classification. It is postulated that 5% of the patients on Roux en Y reconstruction will experience poor clinical symptoms compared to 25% of those on Billroth II based on reflux symptoms. To achieve a statistical significance with 95% power and a 2-sided test of 5% for this 20% clinical difference, 80 subjects for each arm will be required. Factoring a 10% attrition rate for mortality and lost to follow up, a total of 160 subjects to be randomized equally will be recruited.

DETAILED DESCRIPTION:
Subtotal distal gastrectomy with lymphadenectomy offers the best chance of cure either alone or in conjunction with other modalities for patients with operable distal gastric cancer. After a subtotal gastrectomy the gastrointestinal continuity can be restored by various techniques. Billroth I, Billroth II and Roux-en-Y reconstruction are all acceptable procedure with each having its merits and demerits. The choice of reconstructive procedure varies depending on individual Surgeons preference and institutional practice. There is geographical difference in practice with majority of surgeons in the east favoring Billroth I, while in the west; Roux-en-Y is more commonly employed (1). Billroth I vs Roux-en-Y reconstruction has been extensively studied with a prospective series by Sounya Nunobe et al that reported superior symptomatic and functional outcomes of Roux-en-Y procedure (2). However a randomised trial by Makoto Ishikawa et al found limited advantages of Roux-en-Y over Billroth I reconstruction (3). In this study Roux-en-Y had fewer problems related to reflux of bile but a higher incidence of stasis in the Roux limb resulting in longer hospital stay. Another reason that some surgeon avoids doing Roux-en-Y is a triad of post operative symptoms including abdominal pain, vomiting and nausea called Roux-en-Y loop syndrome (4,5). Billroth II reconstruction in comparison to Roux-en-Y is a simpler operation with only one anastomosis and faster operating time (6). This has implications while managing gastric cancer patients who may be malnourished and a simpler procedure may have lesser risk of complications and yield better outcomes. Billroth II has been criticized for increased reflux associated problem like esophagitis and gastritis, also noteworthy are risk of afferent loop and dumping syndrome. Long term nutritional outcomes are similar for both procedures (7).

ELIGIBILITY:
Inclusion Criteria:

* Patient able to give informed consent
* Age 21 - 80 years both male & females
* Patients with histopathologically confirmed adenocarcinoma of the distal lesser curve, distal greater curve, incisura and antrum that are deemed suitable for elective radical subtotal gastrectomy with curative intent.

Exclusion Criteria:

* Unable to give informed consent
* Patients who have undergone previous gastrectomy
* Patients with stomach cancer or previous small bowel surgery precluding construction of either form of anastomosis thus preventing randomization.
* Patients operated for palliation of gastric outlet obstruction, bleeding, perforation and obstruction
* Emergency gastrectomy for complications related to tumor.
* Patients with early gastric cancer who can have curative treatment by endoscopic methods.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-10-09 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to compare Billroth II and Roux En Y reconstruction after radical distal subtotal gastrectomy for gastric cancer in terms of postoperative outcomes. | 1 year
  The outcomes include postoperative gastrointestinal symptoms, nutritional status, gastritis and/or esophagitis on endoscopy and quality of life up to one year after surgery. With the results, we can have a scientific basis in choosing the more suitable method of reconstruction for our patients.

SECONDARY OUTCOMES:
Quality of life pre and post operatively will be compared between Billroth II and Roux En Y reconstruction after radical distal subtotal gastrectomy. | 1 year
  Symptomatic outcomes of both procedures have significant bearing on quality of life of patients and at the end be able to identify the better among the two procedure.
Gastrointestinal symptoms assessment | 1 year
  Grading of clinical symptom is based on the total score of the the five items epigastric pain, heartburn, vomiting bile, postprandial bloating and nausea)pre and post operatively at 1 year. The higher the grade the poorer the outcome.
Assessing nutritional status | 1 year
  Biochemical parameters as well as the height and weight of patients are measured pre operatively, 6 months and 1 year post operatively to compute the BMI. The nutrition assessment are scored by using the NRI and total lymphocyte count.
Grading of gastritis and/or esophagitis on endoscopy | 1 year
  Endoscopic classification of inflammation of the remnant stomach to be graded one year after surgery. The gastritis will be reported according to the updated Sydney classification with the morphologic pattern, etiology & topography being reported.

CONTACTS AND LOCATIONS:
Overall Officials: Asim Shabbir, MBBS, Principal Investigator — National University Hospital System
Locations (4):
- The Chinese University of Hong Kong, Hong Kong, Shatin, NT, Hong Kong
- Singapore (3):
  - National University Hospital, Kent Ridge
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore

REFERENCES:
- [Background] Woodward A, Sillin LF, Wojtowycz AR, Bortoff A. Gastric stasis of solids after Roux gastrectomy: is the jejunal transection important? J Surg Res. 1993 Sep;55(3):317-22. doi: 10.1006/jsre.1993.1148. PMID 8412117
- [Background] Mathias JR, Fernandez A, Sninsky CA, Clench MH, Davis RH. Nausea, vomiting, and abdominal pain after Roux-en-Y anastomosis: motility of the jejunal limb. Gastroenterology. 1985 Jan;88(1 Pt 1):101-7. doi: 10.1016/s0016-5085(85)80140-2. PMID 3964759
- [Background] Yoshino K. [History of gastric cancer surgery]. Nihon Geka Gakkai Zasshi. 2000 Dec;101(12):855-60. Japanese. PMID 11201113
- [Background] Fukuhara K, Osugi H, Takada N, Takemura M, Higashino M, Kinoshita H. Reconstructive procedure after distal gastrectomy for gastric cancer that best prevents duodenogastroesophageal reflux. World J Surg. 2002 Dec;26(12):1452-7. doi: 10.1007/s00268-002-6363-z. Epub 2002 Oct 10. PMID 12370787
- [Result] Osugi H, Fukuhara K, Takada N, Takemura M, Kinoshita H. Reconstructive procedure after distal gastrectomy to prevent remnant gastritis. Hepatogastroenterology. 2004 Jul-Aug;51(58):1215-8. PMID 15239282
- [Result] Nunobe S, Okaro A, Sasako M, Saka M, Fukagawa T, Katai H, Sano T. Billroth 1 versus Roux-en-Y reconstructions: a quality-of-life survey at 5 years. Int J Clin Oncol. 2007 Dec;12(6):433-9. doi: 10.1007/s10147-007-0706-6. Epub 2007 Dec 21. PMID 18071862
- [Result] Ishikawa M, Kitayama J, Kaizaki S, Nakayama H, Ishigami H, Fujii S, Suzuki H, Inoue T, Sako A, Asakage M, Yamashita H, Hatono K, Nagawa H. Prospective randomized trial comparing Billroth I and Roux-en-Y procedures after distal gastrectomy for gastric carcinoma. World J Surg. 2005 Nov;29(11):1415-20; discussion 1421. doi: 10.1007/s00268-005-7830-0. PMID 16240061